CLINICAL TRIAL: NCT03945045
Title: A Randomized Observational Study of the Internal Jugular Vein or the Subclavian Vein Approach for Ultrasound-guided Implantation of Totally Implantable Vascular Access Device(TIVAD)
Brief Title: A Study of the IJV or the SCV Approach for Ultrasound-guided Implantation of TIVAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201807144RINC
Record Dates: First submitted 2019-05-05; First posted 2019-05-10 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Venous Thrombosis; Catheter-Related Infections; Catheter Mechanical Failure Rate
Keywords: venous thrombosis
MeSH Terms: conditions — Venous Thrombosis; Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCV (Experimental): TIVAD implanted through subclavian vein under real-time ultrasound guidance
  Interventions: Procedure: Subclavian vein approach
- IJV (Experimental): TIVAD implanted through internal jugular vein under real-time ultrasound guidance
  Interventions: Procedure: internal jugular vein approach

INTERVENTIONS:
Procedure: Subclavian vein approach — Subclavian vein approach for Ultrasound-guided Implantation of TIVAD
  Other Names: SCV
  Arms: SCV
Procedure: internal jugular vein approach — internal jugular vein approach for Ultrasound-guided Implantation of TIVAD
  Other Names: IJV
  Arms: IJV

SUMMARY:
To compare IJV and SCV as the implantation site of TIVAD and its associated thrombotic or occlusion rate, our study plans to enroll 240 patients with cancer who require central line TIVADs and randomizes them with 1:1 ratio to receive the TIVAD implantation at SCV or IJV. After the implantation, the patients will be regularly followed through phone contact and chart review for 2 years, and any symptomatic thrombosis or occlusion will be found during chemotherapy injection or regular push-pull heparin saline flush every 6 weeks as our hospital care protocol. To detect any asymptomatic thrombosis, the patients will also receive screening vascular ultrasound at 2 weeks, 2 months, and 6 months postoperatively. The study primary endpoints include any infection, asymptomatic thrombosis found by screen ultrasound, and clinically symptomatic thrombosis or occlusion and major mechanical failure/dislocation of TIVAD.

DETAILED DESCRIPTION:
A totally implantable venous access device (TIVAD) provides reliable, long-term vascular access and improves cancer patients' quality of life. The use of TIVADs is associated with important complications as infection and venous thrombosis, and studies have shown that several factors are associated, such as cancer types, catheter types, and the location of the catheter tips. Whether subclavian vein(SCV)or internal jugular vein(IJV) is a better site for TIVAD percutaneous access were also widely studied, and there is no definite consensus generated yet.

A meta-analysis published in 2016 by Wu et al reviewed 12 studies comparing the internal jugular vein (IJV) with the subclavian vein (SCV) as the percutaneous access site found no differences of TIVAD-related infection and catheter-related thrombotic rate. In the secondary outcome, IJV was associated with reduced risks of total major mechanical complications such as catheter dislocation and malfunction. Of 12 studies included, only 3 were randomized trial and there was no consistency between groups of using ultrasound guidance throughout TIVAD insertion. To be further, there is no description of how close to IJV-SCV junction does IJV group were inserted. Hence, a large well-designed RCT is warranted before the IJV site can be recommended.

To compare IJV and SCV as the implantation site of TIVAD and its associated thrombotic or occlusion rate, our study plans to enroll 240 patients with cancer who require central line TIVADs and randomizes them with 1:1 ratio to receive the TIVAD implantation at SCV or IJV. After the implantation, the patients will be regularly followed through phone contact and chart review for 2 years, and any symptomatic thrombosis or occlusion will be found during chemotherapy injection or regular push-pull heparin saline flush every 6 weeks as our hospital care protocol. To detect any asymptomatic thrombosis, the patients will also receive screening vascular ultrasound at 2 weeks, 2 months, and 6 months postoperatively. The study primary endpoints include any infection, asymptomatic thrombosis found by screen ultrasound, and clinically symptomatic thrombosis or occlusion and major mechanical failure/dislocation of TIVAD.

ELIGIBILITY:
Inclusion: 240 cancer patients, 20~99 years old.

Exclusion:

1. Breast cancer, mediastinal tumor above 6 cm, head and neck cancer with/without surgical/radiological treatment, lung tumor above 6 cm,
2. ECOG (Eastern Cooperative Oncology Group)performance status>=2, can't tolerate sit-upright or standing postoperative chest plain film,
3. Allergy to prophylactic antibiotic,
4. History of previous TIVAD or Hickman catheter implantation. Recent 2 weeks Central venous catheter insertion.
5. End stage renal disease.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
infection (blood stream or local wound) | 2 years
  1. catheter-related blood stream infection(CRBSI) due to TIVAD, including:
     1-1. at least one positive blood culture obtained from a peripheral vein, clinical manifestations of infections (i.e., fever, chills, and/or hypotension), and no apparent source for the blood stream infection, except the TIVAD, which leads to the TIVAD removal. Subsequent TIVAD catheter tip culture yields the same organism.
     1-2. Differential time to positivity, with blood culture drawn from the TIVAD that becomes positive at least 2 hr earlier than the peripheral blood culture.
  2. TIVAD local wound infection and/or non-healing will be classified as infection.
asymptomatic venous thrombosis | 2 years
  1. asymptomatic venous thrombosis found by study initiated screening ultrasound at 2 weeks, 2 months, and 6 months postoperatively.
  2. asymptomatic venous thrombosis found by chart review of chest CT/plain film, if exams are available due to other medical indication within 2 years postoperatively.
symptomatic venous thrombosis with positive confirmatory image tests | 2 years
  both positive symptoms and positive confirmative image tests should be met.
  Positive symptom noted by the patient or caregiver, such as
  1. any arm swelling or swelling sensation
  2. suspicious pulmonary embolism with symptom as dyspnea, chest tightness/pain, Hemoptysis...etc.
  Positive confirmatory image tests as
  1. vascular sonography
  2. Catheter-based angiography
  3. Computed tomographic pulmonary angiography (CTPA) or magnetic resonance pulmonary angiography (MRPA)
  4. Ventilation perfusion (V/Q) scanning when pulmonary embolism is suspected.
TIVAD catheter occlusion | 2 years
  Failure or difficult to infuse fluid or withdraw blood from TIVAD. Difficult to withdraw blood from TIVAD in certain body position is not counted.
major mechanical failure, dislocation of TIVAD. | 2 years
  1. catheter kinking, looping, migration to different vessel
  2. catheter disintegration from port.

SECONDARY OUTCOMES:
Intolerable pain or foreign body sensation of TIVAD | 2 years
  1. Subjectively, intolerable "pain or foreign body sensation" of TIVAD, which leads to TIVAD remove without other medical reasons.
  2. Patient requests for TIVAD remove with no pain, no foreign body sensation, and no other medical reasons will not be included in the measure. (that is, "I want to remove TIVAD because TIVAD is an implant")

CONTACTS AND LOCATIONS:
Overall Officials: CHENG-YUAN HSIEH, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan